CLINICAL TRIAL: NCT05005624
Title: Validation of an Activities-of-daily-living Framework at Different Combinations of Light Temperature and Light Intensity
Brief Title: Validation of an Activities-of-daily-living Framework at Different Light Conditions
Status: Completed | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Professor (Associate) of Democritus University of Thrace, Democritus University of Thrace
Other Study IDs: DUTH/EHDE9/29-5-2020
Record Dates: First submitted 2021-08-10; First posted 2021-08-13 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Presbyopia; Near Vision; Reading; Daily Activities
Keywords: activities of daily living; presbyopia; light temperature; light intensity
MeSH Terms: conditions — Presbyopia; Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Validation group 1 (VG-1): 20 participants with binocular Uncorrected Near Visual Acuity (UNVA) 0.1 logMAR (Snellen 20/25)
  Interventions: Other: ADL performance
- Validation group 2 (VG-2): 20 participants with binocular Uncorrected Near Visual Acuity (UNVA) 0.4 logMAR (Snellen 20/50)
  Interventions: Other: ADL performance
- Validation group 3 (VG-3): 20 participants with binocular Uncorrected Near Visual Acuity (UNVA) 0.7 logMAR (Snellen 20/100)
  Interventions: Other: ADL performance

INTERVENTIONS:
Other: ADL performance — All validation groups address the following ten ADL tasks in 9 different combinations of light temperature (in Kelvins - K) and light intensity (in foot candles - fc) in order possible differences to be revealed among the validation groups and light combinations:
  1. Phone Book Search (PBS), 2. Supermarket receipt (SupRe), 3. Book reading (BR), 4. Cellular message (CM), 5. Cellular entry search (CES), 6. Reading computer screen (RCS), 7. Drops bottle reading (DR), 8. Subtitles reading (SubRe), 9. Open door test (ODT), and, 10. Screwdriver test (ST).
  The 9 light combinations are the following:
  3000 K - 25 fc, 3000 K - 50 fc, 3000 K - 75 fc 4000 K - 25 fc, 4000 K - 50 fc, 4000 K - 75 fc 6000 K - 25 fc, 6000 K - 50 fc, 6000 K - 75 fc

SUMMARY:
Primary objective of this study is the construction and validation of an experimental environment for the simulation of a variety of near- and intermediate-vision activities of daily living (ADLs) in different combinations of light temperature and light intensity.

DETAILED DESCRIPTION:
Among the objectives of the study is to validate a framework of ADLs that require near and intermediate vision and better reflect visual capacity, in a special experimental environment of 9 different combinations of light temperature and light intensity.

The final list consists of the following ten basic ADL tasks:

1. Phone Book Search (PBS), 2. Supermarket receipt (SupRe), 3. Book reading (BR), 4. Cellular message (CM), 5. Cellular entry search (CES), 6. Reading computer screen (RCS), 7. Drops bottle reading (DR), 8. Subtitles reading (SubRe), 9. Open door test (ODT), and, 10. Screwdriver test (ST).

The 9 light combinations are the following:

3000 K - 25 fc, 3000 K - 50 fc, 3000 K - 75 fc 4000 K - 25 fc, 4000 K - 50 fc, 4000 K - 75 fc 6000 K - 25 fc, 6000 K - 50 fc, 6000 K - 75 fc

ELIGIBILITY:
Inclusion Criteria:

* normophakic participants with a clear natural lens
* age between 40 to 75 years old
* UNVA: logMAR 0.1, 0.4, or 0.7

Exclusion Criteria:

* astigmatism >1.00 diopters
* glaucoma
* intraocular pressure lowering medications
* former incisional eye surgery
* corneal or fundus disease
* diabetes mellitus
* autoimmune diseases
* neurological, psychiatric or mental diseases

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normophakic participants with a clear natural lens
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Phone Book Search (PBS) score | through study completion, an average of 6 months
  Patient is required to find and read a specific entry in a regular phonebook catalog in the nine different combinations of light temperature and light intensity. A different entry is asked to be found in each combination.
  [scale's best value: 100, scale's worst value: 0]
Supermarket Receipt (SupRe) score | through study completion, an average of 6 months
  Patient is required to find and read three products from a typical supermarket receipt in the nine different combinations of light temperature and light intensity. Different products are asked to be found in each combination.
  [scale's best value: 100, scale's worst value: 0]
Book Reading (BR) score | through study completion, an average of 6 months
  Patient is required to read an excerpt of a predetermined length in a novel in the nine different combinations of light temperature and light intensity. A different excerpt of the same length is asked to be read in each combination.
  [scale's best value: 100, scale's worst value: 0]
Cellular message (CM) score | through study completion, an average of 6 months
  Patient is required to read a Short Message Service (SMS) on a cellular phone in the nine different combinations of light temperature and light intensity. A different SMS is asked to be read in each combination.
  [scale's best value: 100, scale's worst value: 0]
Cellular Entry Search (CES) score | through study completion, an average of 6 months
  Patient is required to find and read one specific entry on a cellular phone in the nine different combinations of light temperature and light intensity. Different entries are asked to be found in each combination.
  [scale's best value: 100, scale's worst value: 0]
Reading Computer Screen (RCS) score | through study completion, an average of 6 months
  Patient is required to correctly read text of a predetermined length from a computer screen in the nine different combinations of light temperature and light intensity. Different texts of the same length are asked to be read in each combination.
  [scale's best value: 100, scale's worst value: 0]
Drops bottle Reading (DR) score | through study completion, an average of 6 months
  Patient is required to correctly read the expiration date printed on three typical eye dropper bottles in the nine different combinations of light temperature and light intensity. Different eye dropper bottles are given to be read in each combination.
  [scale's best value: 100, scale's worst value: 0]
Subtitles Reading (SubRe) score | through study completion, an average of 6 months
  Patient is required to correctly read movie subtitles from a one-minute movie excerpt on a computer screen in the nine different combinations of light temperature and light intensity. Different movie excerpts are shown in each combination.
  [scale's best value: 100, scale's worst value: 0]
Open Door Test (ODT) score | through study completion, an average of 6 months
  Patient is required to find a specific key from a keychain that holds 10 keys and put it in the corresponding door keyhole in the nine different combinations of light temperature and light intensity. Different keychains are given in each combination.
  [scale's best value: 100, scale's worst value: 0]
Screwdriver Test (ST) score | through study completion, an average of 6 months
  Patient is required to select one among three screwdrivers and insert it in the appropriate screw among a variety of screw types in the nine different combinations of light temperature and light intensity. Different screwdrivers are given to be selected in each combination.
  [scale's best value: 100, scale's worst value: 0]

SECONDARY OUTCOMES:
Uncorrected Distance Visual Acuity (UDVA) | through study completion, an average of 6 months
  Monocular and binocular UDVA of all groups is estimated using the Greek version of the Early Treatment Diabetic Retinopathy Study Chart at four meters distance
Uncorrected Intermediate Visual Acuity (UIVA) | through study completion, an average of 6 months
  Monocular and binocular UIVA of all groups is estimated using web-based Democritus Digital Acuity Reading Test (wDDART)
Uncorrected Near Visual Acuity (UNVA) | through study completion, an average of 6 months
  Monocular and binocular UNVA of all groups is estimated using web-based Democritus Digital Acuity Reading Test (wDDART)
25-item National Eye Institute Visual Function Questionnaire (NEI VFQ-25) score | through study completion, an average of 6 months
  Vision-specific quality of life of all participants is evaluated with the Greek version of NEI VFQ-25, which is handed to the patients prior to their ADL assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD, PhD, Study Chair — Department of Ophthalmology, University Hospital of Alexandroupolis, Alexandroupolis, Greece
Locations (1):
- Department of Ophthalmology, University Hospital of Alexandroupolis, Alexandroupoli, Evros, Greece